CLINICAL TRIAL: NCT04824066
Title: The Role of Wearable Devices in Cardiothoracic Surgery: Predicting and Detecting Early Postoperative Complications
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Chi-Fu Jeffrey Yang, MD, Massachusetts General Hospital
Other Study IDs: 2020P002984
Record Dates: First submitted 2021-03-11; First posted 2021-04-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Surgery--Complications
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiothoracic Surgery Cohort: Adults patients who are scheduled to undergo cardiothoracic surgery and meet the inclusion and exclusion criteria.
  Interventions: Device: Device: Wearable Device

INTERVENTIONS:
Device: Device: Wearable Device — A Wearable Device will be placed on the wrist of the patient ~30 days prior to the patient's scheduled surgery, removed during the operation, and replaced for ~180 days post-operatively. The device will record activity in terms of steps, sleep quality, heart rate, etc.

SUMMARY:
The overarching goal of this research is to use machine learning analysis of high-resolution data-collected by wearable technology-of cardiothoracic surgical patients to assess recovery and detect complications at their earliest stage

DETAILED DESCRIPTION:
This is a single-center non-randomized prospective cohort study using wearable devices in cardiothoracic surgery patients to detect post-operative complications. Patients undergoing cardiothoracic surgery who meet the inclusion and exclusion criteria will be enrolled consecutively with verbal informed consent from the time this protocol is approved by the IRB until 1,200 subjects are enrolled. At ~30 days preoperatively the subjects will have a wearable device (such as a Fitbit) placed on their wrist and will wear the device until ~180 days post-operatively. This device will wirelessly transmit data regarding activity and sleep quality to a smartphone application for the duration of wear and data will be analyzed by our collaborators at Case Western Reserve University.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older undergoing cardiothoracic surgery that is male or a non-pregnant female and are amenable to using one of the wearable devices of interest (Fitbit, iWatch, Biostrap).
2. Individuals willing to provide informed consent and who have capacity for all study procedures

Exclusion Criteria:

1. Individuals with mental incapacity and/or cognitive impairment that would preclude adequate understanding of, or cooperation with the study protocol.
2. Any pregnant participant.
3. Severe irreversible pulmonary hypertension.
4. Congenital heart disease
5. Chronic renal insufficiency or undergoing chronic renal replacement therapy
6. Liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiothoracic surgery that are amenable to wearing a device of interest and meet the inclusion and exclusion criteria above will be approached for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Early detection of postoperative complications using machine learning analysis of patient biometric data. | Four Years
  Proportion of complications detected by the machine learning algorithm.
Prediction of the quality of postoperative recovery using pre- and intraoperative data. | Four Years
  Proportion of patients whose quality of postoperative recovery is correctly predicted by the machine learning algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Fu Jeffrey Yang, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States